CLINICAL TRIAL: NCT03253367
Title: Phenomics and Genomics in Clozapine Pharmacotherapy: Current, Former and New Clozapine Users
Brief Title: Phenomics and Genomics of Clozapine Pharmacotherapy
Acronym: CLOZIN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jurjen Luykx (Other)
Responsible Party: Sponsor-Investigator, Jurjen Luykx, Sponsor, UMC Utrecht
Organization: UMC Utrecht (Other)
Other Study IDs: ABR: 52726 & 52728
Record Dates: First submitted 2017-05-29; First posted 2017-08-17 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Schizophrenia Spectrum and Other Psychotic Disorders
Keywords: Schizophrenia Spectrum and Other Psychotic Disorders
MeSH Terms: conditions — Schizophrenia Spectrum and Other Psychotic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — For current and former users we obtain DNA and for new users we also obtain RNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Current/former clozapine users: This group has only one visit.
  Interventions: Other: Blood is obtained, mostly during routine venipuncture
- New clozapine users: This group will be followed for 6 months prospectively.
  Interventions: Other: Blood is obtained, mostly during routine venipuncture

INTERVENTIONS:
Other: Blood is obtained, mostly during routine venipuncture

SUMMARY:
A burgeoning body of research has pointed to increased efficacy of clozapine (CLZ) over other antipsychotics in schizophrenia (SCZ). On the other hand, safety concerns likely cause underutilization across a range of European and other nations. The lack of data available to predict efficacy and adverse drug reactions (ADRs) of CLZ further contributes to underprescription rates in these countries. Here, we hypothesize that (epi)genetic and non-genetic factors aid to help predict treatment outcome (efficacy + ADRs) to CLZ. We furthermore posit that such prediction will result in enhanced quality of life of both patients and family members. Our primary objective is to predict CLZ treatment outcome based on phenotypic and genetic data obtained through the current design. The first secondary objective is to investigate which methylation levels/patterns are correlated with CLZ treatment outcome. The second secondary objective is to aid in the further elucidation of the genetic architecture of SCZ and any possible differences between 'regular' SCZ patients and those on CLZ, who are generally more severely ill. We thus intend to cover two currently unmet needs using a precision medicine approach: the lack of knowledge about determinants of treatment response to CLZ and the lack of insight into neurobiological differences between 'regular' SCZ and relatively treatment resistant subjects (CLZ users). The prime analysis will be a common variant hypothesis-generating genotyping endeavor investigating treatment response to CLZ. Additional analyses include whole-genome methylation and gene expression analyses and analyses of non-genetic determinants of response. We will include 2,500 CLZ treated patients for our discovery cohort, which is in line with previous whole-genome pharmacogenomics studies and our power calculations. We will replicate any genome-wide loci using our prospectively collected cohort of new users (N=59). Potential yields include a publicly available prediction tool to help identify patients responsive to CLZ in early disease stages and prevent harmful effects. In addition, common variant analyses compounded by pathway analyses may help elucidate the mechanisms of action of CLZ. We ask for broad informed consent from participants ensuring rich, longitudinal phenotypic and genotypic data resources for both currently planned and future analyses, allowing e.g. next-generation sequencing focused on both CLZ and SCZ disease genetics (e.g. in large consortia). We plan to also generate polygenic risk scores (PRS) of CLZ efficacy and use those to identify other diseases or patients for which CLZ may be helpful, e.g. schizoaffective disorder patients who are sometimes first treated with mood stabilizers. Last, evidence hints that disparaging genetic loci influence efficacy to different antipsychotics. Adding genetic data from our cohort to existing datasets of response to other antipsychotics may help identify such loci. Finally, comparison studies with non-CLZ using patients suffering from SCZ may deepen the understanding of biological mechanisms underlying treatment resistance (or: a relatively severe course of illness).The results of this genetic part of the study will be combined with the results from our other research protocol 'Phenomics and genomic of clozapine pharmacotherapy - New Users'.The overarching goal of both projects is to create a prediction model for clozapine outcome (response (and side effects). This model includes genetic, epigenetic and clinical data.

DETAILED DESCRIPTION:
Rationale Clozapine (CLZ) is generally prescribed if at least two trials of antipsychotic agents have not led to satisfactory clinical improvement, thereby implying that patients on CLZ generally suffer from more severe and/or persistent symptoms than patients suffering from schizophrenia spectrum disorders (SCZ) on other antipsychotic agents. Unraveling the (functional) genetic variation underlying this severe SCZ phenotype therefore has the potential to deepen our understanding of the biological underpinnings of SCZ beyond the boundaries of DSM-based consensus criteria. Such knowledge in turn has the potential to shape future pharmacotherapeutic research. The investigators here hypothesize that targeting this phenotype in genome-wide association studies and next-generation sequencing studies will signal genetic risk loci implicated in this severe SCZ phenotype. In the future, this may lead to early detection of severe SCZ, which in turn will enable tailoring of pharmacotherapeutic strategies to such SCZ subtypes. The results of this genetic part of the study will be combined with the results from our other research protocol ('Phenomics and genomic of clozapine pharmacotherapy - New Users').The overarching goal of both projects is to create a prediction model for clozapine outcome (response (and side effects). This model includes genetic, epigenetic and clinical data.

Objectives

Primary:

1) To predict CLZ efficacy and ADRs (=treatment outcome) based on phenotypic and genetic data obtained in this study.

Secondary:

1. To investigate which non-genetic factors, methylation and gene expression levels/patterns predict treatment outcome after initiating CLZ;
2. As the genetic architecture of SCZ has not been fully elucidated, the current project will aid in the further elucidation of the genetic architecture of SCZ and any possible differences between 'regular' SCZ patients (those not considered treatment resistant) and those on CLZ (considered generally to be a more homogeneous and severe group).

Study design This is a mostly cross-sectional study, in which both phenotypic and genotypic data are gathered from this study population that currently uses CLZ or has used CLZ in the past. A genome-wide association study (GWAS) will be performed to reveal possible differences in genetic architecture between patients who use or have used CLZ and the broad schizophrenia phenotype on the one hand and between those who use or have used CLZ and healthy controls on the other. Targeted next-generation sequencing may be used to follow-up possible positive associations. The genetic data will be used to analyse which genetic variants are associated with CLZ response and/or side effects.

Study population The investigators will include 2,500 patients diagnosed with schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder NOS (together referred to as SCZ) >18 years of age who are currently on CLZ treatment or have used CLZ in the past. Publicly available Psychiatric Genomics Consortium (PGC) GWAS data will be used for comparisons with the broad schizophrenia phenotype group. For the purpose of the case-control comparison, the 2,500 subjects who use or have used CLZ will be age and sex-matched to 30,000 healthy control subjects for whom genotype data are available in-house.

Intervention No intervention will be applied.

Main study parameters/endpoints

1. To assess whether the genetic architecture of this severe SCZ phenotype differs from the broad DSM-based SCZ phenotype.
2. To predict clozapine response and side effects based on phenotypic and genetic data obtained in this study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness Almost all patients on CLZ regularly have their blood drawn for routine white blood cell counts and/or CLZ blood level assessments. The investigators anticipate that the majority of the study population will consist of such patients as white blood cell monitoring is strictly enforced in clinical practice for this patient group. For these patients, no additional risks will be attached to the study, as the blood necessary for DNA extraction for the current study will be drawn during these routinely performed venipunctures. Time investment will also be low as the patients will only undergo a 10-minute interview. A minority of patients on CLZ does not have their blood routinely monitored and neither do patients who have used CLZ in the past. These subjects will be asked to allow a single blood draw. A venipuncture entails the risk of a hematoma (blood leaving the vessel). The investigators aim to minimize this risk by only allowing experienced personnel to draw blood and in the event of deeply located or thin veins request central lab personnel to perform the venipuncture. Although a hematoma resulting from a traumatic puncture imposes an esthetical burden on the subject, no serious health risks are involved.

ELIGIBILITY:
Inclusion Criteria:

* he/she currently uses CLZ or he/she has used CLZ in the past/will use CLZ
* he/she has received a diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder NOS.
* his/her age must be ≥18 years old
* he/she must be able to speak and read the language of the Informed Consent (differs per country)
* he/she must be mentally competent and have decisional capacity with regard to a decision to participate in the current study

Exclusion Criteria:

* admission to a psychiatric unit involuntarily (not all countries)
* a history of Parkinson's disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include 2,500 patients diagnosed with schizophrenia, schizophreniform disorder, schizoaffective disorder or psychotic disorder NOS (together referred to as SCZ) >18 years of age who are currently on CLZ treatment or have used CLZ in the past. Publicly available Psychiatric Genomics Consortium (PGC) GWAS data will be used for comparisons with the broad schizophrenia phenotype group. For the purpose of the case-control comparison, the 2,500 subjects who use or have used CLZ will be age and sex-matched to 13,000 healthy control subjects for whom genotype data are available in-house.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2016-01-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Predict clozapine response. | 2016-2021
  To predict clozapine response based on phenotypic information from our questionnaire (CGI + CRES) and genetic information from GWAS
Predict side effects from clozapine use | 2016-2021
  To predict clozapine response based on phenotypic information from our questionnaire (LUNSERS) and genetic information from GWAS
Assess differences in genetic architecture (GWAS) | 2016-2021
  To assess whether the genetic architecture of this severe SCZ phenotype differs from the broad DSM-based SCZ phenotype. this will be done by comparing the gentic material of clozapine users vs. non-clozapine users. Only the clozapine DNA has to be collected yet.

SECONDARY OUTCOMES:
Detect genetic associations (GWAS) Detect genetic associations current severe SCZ phenotype | 2016-2021
  To detect genetic associations with the current severe SCZ phenotype by performing a case-control comparison with healthy participants (GWAS).
Increase or decrease cardiovascular disease? | 2016-2031
  To investigate whether CLZ use increases or decreases the risk of cardiovascular disease and early death. This is done by following the patients for 10 years and see whether they developed serious cardiovascular diseases

CONTACTS AND LOCATIONS:
Locations (11):
- Medical University Innsbruck, Innsbruck, Austria
- Niuvanniemen hospital, Kuopio, Finland
- Germany (2):
  - LMU Munich, München, Munich
  - Charité Universitätsmedizin Berlin, Berlin
- Netherlands (7):
  - Vincent van Gogh Institute, Venray, Limburg
  - Reinier van Arkel, 's-Hertogenbosch, North Brabant
  - GGZ-NHN, Heerhugowaard, North Holland
  - GGZ Rivierduinen, Leiden, Oegstgeest
  - Yulius, Barendrecht, South Holland
  - UMC Utrecht, Utrecht
  - Altrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Yes
Anonymous data can be shared with other investigators when the sponsor agreed on the workpackage of that investigator.

REFERENCES:
- See also: Website CLOZIN study — http://www.clozinstudy.com